CLINICAL TRIAL: NCT02724813
Title: Tele-rehabilitation for Cognitive Disability Post Stroke: Enhancing Function in the Face of Geographical Disparities
Brief Title: Tele-Rehabilitation Study for People With a History of Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Collaborators: Health and Stroke Foundation-Canadian Partnership for Stroke recovery (Unknown)
Responsible Party: Principal Investigator, Dr. Deirdre Dawson, Senior Scientist, Baycrest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB#15-37
Record Dates: First submitted 2016-02-09; First posted 2016-03-31 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm (Experimental): Participants will receive 16 one-hour tele-CO-OP sessions delivered over a 10-week period by a licensed health care professional. We will deliver tele-CO-OP via Skype™ and record all sessions using Pamela software for Skype™.
  Interventions: Behavioral: Cognitive Orientation to Occupational Preformance (COOP)
- Wait-list arm (Active Comparator): Participant in this arm will receive therapy 8 weeks after initial assessment. Participants will receive 16 one-hour tele-CO-OP sessions delivered over a 10-week period by a licensed health care professional. We will deliver tele-CO-OP via Skype™ and record all sessions using Pamela software for Skype™.
  Interventions: Behavioral: Cognitive Orientation to Occupational Preformance (COOP)

INTERVENTIONS:
Behavioral: Cognitive Orientation to Occupational Preformance (COOP)

SUMMARY:
Stroke results in long-term disability for many people, and particularly for survivors of stroke who have cognitive impairments. However, a decreasing proportion of stroke patients are able to access or receive publicly funded rehabilitation. The investigators have shown in previous studies that in-person delivery of the Cognitive Orientation to daily Occupational Performance (CO-OP) rehabilitation approach to promoting attainment of everyday life goals has resulted in improvements in functional independence and executive function. In a small pilot study of tele-CO-OP with people with chronic traumatic brain injury (TBI) (n=3), the investigators found the delivery method was feasible and that participants were satisfied with the treatment and demonstrated clinically significant improvements on personally meaningful activities. The investigators will investigate the feasibility, preliminary efficacy, and cost-effectiveness of delivering CO-OP in an online format to reduce disability post-stroke. The study design is a single-blind (assessor), randomized wait-list control trial with a one-month retention follow-up. All therapy and testing sessions will be delivered online. We hypothesize that participants will demonstrate improvement in everyday activities and community participation.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults at least three months post-stroke
* Fluent in written and spoken English
* Impairment of executive cognitive functions
* Ability to self-identify specific areas of difficulty in their everyday life that they would like to improve
* Access to a computer or tablet with a high-speed internet connection

Exclusion Criteria:

* Presence of dementia
* Severe concurrent depression
* Severe aphasia
* Concurrent substance abuse

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-09-30 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in Canadian Occupational Performance Measure (COPM) | 10 weeks and 14 weeks
  The COPM is a standardized, semi-structured interview that facilitates goal identification and has been used as the primary outcome measure for many of the CO-OP studies
Changes in Reintegration to Normal Living Index (RNL) | 10 weeks and 14 weeks
  The RNL is a measure of satisfaction with participation in everyday life

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Dawson, PhD, Principal Investigator — Baycrest Health Sciences
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dawson DR, Anderson ND, Binns M, Bar Y, Chui A, Gill N, Linkewich E, McEwen S, Nalder E, Skidmore E. Strategy-training post-stroke via tele-rehabilitation: a pilot randomized controlled trial. Disabil Rehabil. 2024 Jan;46(1):67-76. doi: 10.1080/09638288.2022.2154397. Epub 2022 Dec 14. PMID 36524387